CLINICAL TRIAL: NCT03283345
Title: ASSESSMENT OF SYSTEMIC RESPONSES TO TRAUMA IN DIFFERENT PHASES OF THE MENSTRUAL CYCLE: IN PATIENTS UNDERWENT MODIFIED RADICAL MASTECTOMY A Clinical Study
Brief Title: Effect of Menstrual Cycle on Traumatic Systemic Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hayal Uzelli Şimşek, Principal investigator, Kocaeli University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008/69
Record Dates: First submitted 2017-08-20; First posted 2017-09-14 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: breast cancer; menstrual cycle; breast surgery; systemic responses to trauma
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Breast Neoplasms | interventions — Mastectomy, Modified Radical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postmenopausal women (Active Comparator): postmenopausal female breast cancer patients who underwent modified radical mastectomy
  Interventions: Procedure: modified radical mastectomy
- premenopausal women (Active Comparator): premenopausal female breast cancer patients who underwent modified radical mastectomy
  Interventions: Procedure: modified radical mastectomy

INTERVENTIONS:
Procedure: modified radical mastectomy — systemic responses to trauma are compared with evaluating inflammatory cytokine levels between premenopausal and postmenopausal patient groups with different estrogen levels who underwent modified radical mastectomy.

SUMMARY:
It is aimed to evaluate pathophysiology of systemic responses to trauma via using interleukin (IL) -1 and IL-6 levels and determining timing of surgery through phases of menstrual cycle.

DETAILED DESCRIPTION:
89 female breast cancer patient who underwent modified radical mastectomy included into study. Menstrual history and hormone levels were used to determine menstrual phase: luteal, follicular, and other. IL-1β and IL-6 levels, which are related to severeness of inflammation, were measured one day before and one day after surgery. Those are statistically analysed to show effect of timing of breast surgery on responses to trauma in postmenopausal and premenopausal women during different phases of their menstrual cycles

ELIGIBILITY:
Inclusion Criteria:

* female patients
* who underwent modified radical mastectomy for breast cancer
* who signed informed consent forms

Exclusion Criteria:

* For premenopausal patients taking oral contraceptives
* for postmenopausal patients taking hormone replacement therapy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 89 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
IL-1 and IL-6 levels | 5 month
  evaluate pathophysiology of systemic responses to trauma via using IL-1 and IL-6 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Cantürk, Study Director — Kocaeli University